CLINICAL TRIAL: NCT02768649
Title: A Phase I, Open Label, Single Center, Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetic Profile of RBP-7000 at Low, Medium, and High Doses
Brief Title: Single Ascending Dose Study of RBP-7000
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RB-US-09-0008
Record Dates: First submitted 2016-05-03; First posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Eligible subjects received a test dose of 0.25 risperidone prior to dosing with RBP-7000. Fifteen eligible subjects then received low dose RBP-7000
  Interventions: Drug: RBP-7000; Drug: risperidone
- Cohort 2 (Experimental): After safety and tolerability review of the data from Day 1 to Day 15 of the low dose arm, 3 subjects were dosed in Cohort 2 with a higher dose of RBP-7000. A safety and tolerability review of the data from Day 1 to Day 15 was completed for the 3 subjects before the remaining 12 were dosed.
  Interventions: Drug: RBP-7000; Drug: risperidone
- Cohort 3 (Experimental): After safety and tolerability review of the data from Day 1 to Day 15 of the medium dose arm, 3 subjects were dosed in Cohort 3 with a higher dose of RBP-7000. A safety and tolerability review of the data from Day 1 to Day 15 was completed for the 3 subjects before the remaining 12 were dosed.
  Interventions: Drug: RBP-7000; Drug: risperidone

INTERVENTIONS:
Drug: RBP-7000 — Sequential dosing of each cohort
Drug: risperidone — All eligible subjects received a test dose of risperidone to ensure tolerability prior to dosing with RBP-7000.
  Other Names: test dose

SUMMARY:
The purpose of this study was to assess the safety and tolerability of injections of RBP-7000 in subjects with stable schizophrenia

DETAILED DESCRIPTION:
This was an open-label, single-center, Phase 1, single ascending dose study, designed to evaluate the safety, tolerability, and pharmacokinetic (PK) profile of a single SC injection of low, medium and high doses of RBP-7000 in subjects with clinically stable schizophrenia who were not taking risperidone. The design was a sequential cohort with treatment initiated in 3 cohorts after safety and tolerability at a lower dose were confirmed.

Eligible subjects received a single oral test dose of 0.25mg risperidone under medical supervision. Subjects who continued to be eligible were admitted to a residential unit for approximately 14 days, and received a single dose of RBP-7000. Subjects were discharged on Day 15 and returned to the clinical site weekly for approximately 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with confirmed diagnosis of paranoid, residual, or undifferentiated schizophrenia in a documented letter from the subject's psychiatrist or primary care provider.
* Clinically stable subjects (subjects whom the PI established by medical record or by history from the subject and at least 1 reliable informant, that the subject had been clinically stable for at least 60 days without hospitalization).
* Subjects with body mass index (BMI) between 18 and 33 kg/m2 and weight of at least 49.9 kg.
* Subjects who gave written informed consent.

Exclusion Criteria:

* Subjects taking any risperidone product within the last 60 days prior to study screening.
* Subjects with a history of cancer (excluding resected basal cell or squamous cell carcinoma of the skin) unless they had been disease free for ≥ 5 years.
* Subjects with another active medical condition or organ disease that could have either compromised subject safety or interfered with the safety and/or outcome evaluation of the study drug. This included, but was not limited to the following abnormalities: total bilirubin > 2.5 mg/dL (51 μmol/L), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 × the upper limit of normal (ULN) or clinically significant serum creatinine > 2 x ULN, international normalized ratio (INR) ≥ 2.0. Other excluded medical conditions included, but were not limited to: history of heart attack, brain injury, low blood pressure, and clinically significant irregular heartbeat as interpreted by the PI.
* Subjects who were known to have acquired immune deficiency syndrome or to be human immunodeficiency virus (HIV) positive.
* Subjects with evidence or history of significant hepatic disorder, including acute or chronic hepatitis B and acute hepatitis C. Subjects with hepatitis C antibody and liver functions ≤ 1.5 times the ULN could be included in the study.
* Subjects with known diagnosis of type 1 or 2 diabetes or subjects with a clinically significant abnormal hemoglobin A1c (HbA1c) at screening as interpreted by the PI.
* Subjects with clinically significant comorbidities that could affect near-term survival.
* Subjects treated with any investigational drug within the last 30 days prior to study screening.
* Subjects with significant traumatic injury, major surgery, or open biopsy within the last 4 weeks prior to study screening.
* Subjects receiving opioid or opioid-containing analgesics within the last 30 days prior to study screening.
* Subjects consuming > 1 alcoholic drink per day within the last 30 days prior to study screening (defined as 1 oz. of 80 proof spirits, 12 oz. of beer, or 4 oz. of wine).
* Subjects with prior allergic reactions, sensitivities, or other known contraindications to any component of RBP-7000 (i.e., risperidone, poly [DL-lactide-co-glycolide], or N-methylpyrrolidone).
* Subjects with other concurrent uncontrolled illness that may have interfered with the ability to participate in the study.
* Women with a positive pregnancy test at screening. Women of childbearing potential, who were pregnant or lactating, seeking pregnancy, or failing to take adequate contraceptive precautions (e.g., an oral or injectable contraceptive, an approved hormonal implant or topical patch, or an intrauterine device). Should a female subject become sexually active, she must have agreed to use a double-barrier method or barrier plus spermicide. A woman of childbearing potential was defined as any female who was less than 2 years post-menopausal or had not undergone a hysterectomy or surgical sterilization, e.g., bilateral tubal ligation or bilateral ovariectomy (oophorectomy). Females who were post-menopausal were confirmed by the follicle stimulating hormone (FSH) test at initial screening.
* Subjects with a positive urine drug screen for opioids, cocaine, amphetamines, methadone, marijuana, barbiturates, benzodiazepines, methamphetamine, phencyclidine, or tricyclic antidepressants unless the positive screen was determined to be secondary to an allowable concomitant medication.
* Subjects with epilepsy or other seizure disorders, Parkinson's disease, or dementia.
* Subjects taking bupropion, chlorpheniramine, cimetidine, clomipramine, doxepin, or quinidine within the last 30 days prior to study screening.
* Subjects taking clozapine, phenothiazines, aripiprazole, or haloperidol within the last 30 days prior to study screening.
* Subjects taking serotonin reuptake inhibitors (e.g., fluoxetine, paroxetine) within the last 30 days prior to study screening.
* Subjects taking medications, in addition to those listed above, which may have been expected to significantly interfere with the metabolism or excretion of risperidone and/or 9-hydroxyrisperidone that may have been associated with a significant drug interaction with risperidone, or may have posed a significant risk to subjects' participation in the study.
* Subjects who had been previously injected with RBP-7000 in this study. Subjects who were unable, in the opinion of the PI, to comply fully with the study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] after a subcutaneous injection of a single 60 mg, 90 mg, and 120 mg dose of risperidone in RBP-7000 in subjects with clinically stable schizophrenia | Day 1 through Day 85
  Adverse events, serious adverse events, and discontinuations due to AEs related to treatment.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of risperidone and total risperidone | Day 0 through Day 85
  Blood samples for PK were collected and analyzed for concentration data of risperidone, 9-hydroxyrisperidone, and total risperidone throughout the study period
Time of occurrence of Cmax (Tmax) of risperidone and total risperidone | Day 0 through time of last quantifiable concentration
  Blood samples for PK were collected and analyzed for concentration-time data of risperidone, 9-hydroxyrisperidone, and total risperidone throughout the study period
Area under the plasma concentration versus time curve (AUC) | Day 0 through Day 85
  Area under the risperidone and total risperidone plasma concentration-time curves from time-zero to Day 85
Observed terminal rate constant of risperidone and total risperidone (λz) | Day 0 through Day 85
  λz estimated by linear regression through at least 3 data points in the terminal phase of the log concentration-time profile
Terminal half-life of risperidone and total risperidone (T1/2) | Day 0 through Day 85
  The observed terminal half-life of risperidone, 9-hydroxyrisperidone, and total risperidone was calculated

CONTACTS AND LOCATIONS:
Locations (1):
- CRI Worldwide, Willingboro, New Jersey, United States